CLINICAL TRIAL: NCT01867710
Title: A Randomized Phase 2 Study Evaluating Abiraterone Acetate With Different Steroid Regimens for Preventing Symptoms Associated With Mineralocorticoid Excess in Asymptomatic, Chemotherapy-naïve and Metastatic Castration-resistant Prostate Cancer (mCRPC) Patients
Brief Title: Abiraterone With Different Steroid Regimens for Side Effect Related to Mineralcorticoid Excess Prevention in Prostate Cancer Prior to Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR100916; 2012-004331-23 (EudraCT Number); 212082PCR2023 (Other: Janssen CTMS ID)
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Results first posted 2016-05-11 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Prostate Cancer
Keywords: Mineralocorticoid Excess ; Chemotherapy-Naïve; Metastatic Castration-Resistant Prostate Cancer; Abiraterone Acetate; Zytiga; Prednisone; dexamethasone
MeSH Terms: conditions — Prostatic Neoplasms; Hyperaldosteronism | interventions — Abiraterone Acetate; Prednisone; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (4):
- AA + prednisone 5 mg twice daily (Experimental): Abiraterone acetate in combination with prednisone 5 mg twice daily
  Interventions: Drug: Abiraterone Acetate; Drug: Prednisone 5 mg twice daily
- AA + prednisone 5 mg once daily (Experimental): Abiraterone acetate in combination with prednisone 5 mg once daily dose
  Interventions: Drug: Abiraterone Acetate; Drug: Prednisone 5 mg once daily
- AA + prednisone 2.5 mg twice daily (Experimental): Abiraterone acetate in combination with prednisone 2.5 mg twice daily
  Interventions: Drug: Abiraterone Acetate; Drug: Prednisone 2.5 mg twice daily
- AA + dexamethasone 0.5 mg once daily (Experimental): Abiraterone acetate in combination with dexamethasone 0.5 mg once daily
  Interventions: Drug: Abiraterone Acetate; Drug: Dexamethasone 0.5 mg once daily

INTERVENTIONS:
Drug: Abiraterone Acetate — Type = exact number; unit = mg; number = 1000; form = tablet; route = oral; taken as four 250 mg tablets once daily at least 2 hours after eating and no food should be eaten for at least 1 hour after taking the tablets.
Drug: Prednisone 5 mg twice daily — type = exact number; unit = mg; number = 5; form = tablet; route = oral; taken twice daily, the first dose in the morning after a meal and the second dose after a minimum interval of 8 hours in the late afternoon or early evening, after a meal
  Arms: AA + prednisone 5 mg twice daily
Drug: Prednisone 5 mg once daily — type = exact number; unit = mg; number = 5; form = tablet; route = oral; taken once daily, in the morning after a meal
  Arms: AA + prednisone 5 mg once daily
Drug: Prednisone 2.5 mg twice daily — type = exact number; unit = mg; number = 2.5; form = tablet; route = oral; taken twice daily, the first dose in the morning after a meal and the second dose after a minimum interval of 8 hours in the late afternoon or early evening, after a meal
  Arms: AA + prednisone 2.5 mg twice daily
Drug: Dexamethasone 0.5 mg once daily — type = exact number; unit = mg; number = 0.5; form = tablet; route = oral; taken once daily, in the morning after breakfast
  Arms: AA + dexamethasone 0.5 mg once daily

SUMMARY:
The purpose of the study is to determine the safety and clinical benefit of the combinations of abiraterone acetate and prednisone or abiraterone and dexamethasone in prostate cancer patients. Prednisone will be given at one of three different dose schedules. Dexamethasone will be given at one dose schedule. This will include looking at what side effects occur and how often they occur. In addition the impact of the study drug on quality of life and pain will be evaluated. The study will also collect data on subsequent treatment of patients after they come off the study drug (approximately 4.5 years after the start of study treatment of the first subject participating in the study). By analyzing blood samples, the study aims to identify if some markers could help to understand if the treatment with abiraterone is effective and also help to understand if patients can become resistant.

DETAILED DESCRIPTION:
This is a randomized (study drug is assigned by chance), open-label (all people know the identity of the intervention), parallel-arm, multicenter, phase 2 study of treatment with abiraterone acetate (AA) and 4 alternative steroid treatment strategies in asymptomatic, chemotherapy-naïve, mCRPC patients. A target of 144 patients will be enrolled in this study with 36 patients planned per treatment arm. All patients participating in this study will receive abiraterone acetate. All patients will also take either prednisone or dexamethasone. Patients will receive abiraterone acetate along with either prednisone at one of three different dose schedules or with dexamethasone at one dose schedule. Patients may also be asked to take a medication to protect from osteoporosis as this can be increased by long term use of corticosteroids. There are 4 treatment groups in this study: (a) Four 250 mg tablets of abiraterone acetate taken together once daily and one 2.5 mg tablet of prednisone taken twice daily; (b) Four 250 mg tablets of abiraterone acetate taken together once daily and one 5 mg tablet of prednisone taken once daily; (c) Four 250mg tablets of abiraterone acetate taken together once daily and one 5 mg tablet of prednisone taken twice daily; (d) Four 250 mg tablets of abiraterone acetate taken together once daily and one 0.5 mg tablet of dexamethasone taken once daily. The chance that patients will get prednisone is 3 out of 4 patients. The chance that they will get dexamethasone is 1 out of 4 patients. Abiraterone acetate, prednisone and dexamethasone will be considered as study drugs. The main study will consist of a screening phase of 4 weeks followed by an open-label treatment period of a maximum of 39 treatment cycles (156 weeks or approximately 3 years). The main study treatment period cut-off date will be 156 weeks after the start of study treatment for the first patient participating in the study. Patients will participate in the main study treatment period until the cut-off date, and will receive study treatment until radiographic disease progression and/or unequivocal clinical progression and/or other specific reasons for discontinuation of treatment. Patients will be asked if they would be willing to participate in a follow-up or extension phase of the study for approximately 4.5 years after the start of study treatment of the first subject participating in the study. The amount of time patients will be in the study will vary depending when they join the study and time remaining to the study end date and on their response to the treatment. Patients may come off the study drug if their cancer worsens, if they are unable to tolerate the study treatment, if their doctor determines that they should begin another cancer treatment, or if they decide to withdraw consent. A treatment "cycle" in this study is the amount of time a patient will be asked to take the study medication, and have regularly pre-scheduled checkups and laboratory assessments. Each treatment-cycle will last 28 days. There are a maximum of 39 treatment cycles in this study (over a period of 156 weeks). If patients enter the extension phase, they will be asked to attend hospital every 12 weeks for the remaining time that they stay on the study. Other anticancer therapy or immunotherapy must be ended before and while participating in this clinical study with abiraterone acetate. Also some medications are not allowed during the study. For example, if patients are receiving a steroid other than prednisone, it will be necessary to switch it to prednisone or dexamethasone, depending on to which treatment group patients have been assigned, for the duration of the study. If needed, their study doctor may slowly decrease and stop some or all of their current medicines before the study treatment starts. This is called washout. Do not stop taking any of their current medicine unless their study doctor tells patients to do so. At screening the study doctor will first check that patients are qualified. Screening procedures will be conducted within 4 weeks before randomization. During the main study treatment phase patients will come to the study clinic for Study Visits about 21 times in total (including for screening) if they stay on treatment for 39 cycles. During Cycle 1 of this study, patients will be asked to come to the clinic three times for assessments: on Day 1 which also will usually be their first day of treatment, Day 15 and two weeks later. After that patients will need to return to the clinic once every four weeks for the first 6 months. After that, the visits are once every 3 months for assessments. In addition, patients will need to visit either the clinic or the Outpatients every 2 weeks for the first 3 months and every 4 weeks after that to the end of their treatment to provide a small quantity of blood for testing. If patients either continue study treatment to 39 cycles, or if patients discontinue from the study before 39 treatment cycles, their last visit with drug dispensed will be called an End-of-main-study-treatment (EOMT) visit. EOMT assessments will be performed for all patients who started study treatment, either at the cut-off date or when they discontinue before the cut-off date. Additionally, for patients discontinuing study treatment before the cut-off date, an end-of-main-study (EOMS) visit will be performed 4 weeks after study medication is stopped. Patients will also be required to return to the study site 4 weeks after their last treatment for the "End of Main Study" visit as below. This visit is for some routine study assessments. During the extension phase, patients will be provided with study drug outside of the main study for approximately 4.5 years after the start of study treatment of the first subject participating in the study. During this phase, patients will receive study drug during their 12 weekly visits and their doctor will check on their health status at the same time. Patients will not be required to provide blood or urine samples during this phase. Patients are likely to be eligible to join this extension phase if patients have responded well to the study drug and have not been discontinued from the main study. Also even if they have discontinued from the main study, if they have had no disease progression their doctor may advise them that they are eligible to join this phase. Their last visit will be called an End of Extension visit. For this visit, patients will be required to return to the study site 4 weeks after their last treatment for some final assessments. Follow-Up: Following discontinuation of study treatment at any time during the study, for any reason other than withdrawal of consent, survival and subsequent prostate cancer therapies will be monitored approximately 4.5 years after the start of study treatment of the first subject participating in the study. This information will be obtained by 6-monthly telephone contact and/or chart review, with a source data verification visit scheduled after the death of the patient or at the end of the study. Their doctor may phone them or their family to ask about their health status during this approximately 4.5 years of period if he/she feels that their chart records may need to be updated. A Scientific Advisory Committee will be commissioned to ensure scientific validity of this study, to identify any scientifically relevant trends, and to provide recommendations to the sponsor.

ELIGIBILITY:
Inclusion Criteria:

Have a histologically or cytologically confirmed adenocarcinoma of the prostate Have metastatic disease documented by positive bone scan or by computed tomography or magnetic resonance imaging Have prostate cancer progression documented by prostate specific antigen according to Prostate Cancer Working Group 2 or radiographic progression according to modified RECIST (response evaluation criteria in solid tumors, v1.1) criteria Be asymptomatic from prostate cancer. A score of 0-1 on BPI-SF Question #3 (worst pain in last 24 hours) will be considered asymptomatic Be surgically or medically castrated, with testosterone levels of <50 ng/dL (<2.0 nmol/L). If the subject is being treated with luteinizing hormone releasing hormone (LHRH) agonists or antagonists (subjects who have not undergone orchiectomy), this therapy must have been initiated at least 4 weeks prior to Day 1, Cycle 1 and must be continued throughout the study.

Exclusion Criteria:

Has a history of pituitary or adrenal dysfunction Has an active infection or other medical condition that would contraindicate corticosteroid use Has any chronic medical condition requiring corticosteroid treatment or has received prior corticosteroid treatment for prostate cancer Has a pathological finding consistent with small cell carcinoma of the prostate Has a known brain metastasis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2013-07-16 (Actual); Primary Completion 2015-04-20 (Actual); Study Completion 2018-06-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- Belgium (6):
  - Aalst
  - Brussels
  - Ghent
  - Hasselt
  - Kortrijk
  - Leuven
- Germany (4):
  - Hanover
  - Mülheim
  - Nürtingen
  - Tübingen
- Hungary (2):
  - Budapest
  - Miskolc
- United Kingdom (5):
  - Birmingham
  - Glasgow
  - London
  - Sutton
  - Whitchurch

REFERENCES:
- [Derived] Jayaram A, Wingate A, Wetterskog D, Wheeler G, Sternberg CN, Jones R, Berruti A, Lefresne F, Lahaye M, Thomas S, Gormley M, Meacham F, Garg K, Lim LP, Merseburger AS, Tombal B, Ricci D, Attard G. Plasma tumor gene conversions after one cycle abiraterone acetate for metastatic castration-resistant prostate cancer: a biomarker analysis of a multicenter international trial. Ann Oncol. 2021 Jun;32(6):726-735. doi: 10.1016/j.annonc.2021.03.196. Epub 2021 Mar 29. PMID 33794293
- [Derived] Jayaram A, Wingate A, Wetterskog D, Conteduca V, Khalaf D, Sharabiani MTA, Calabro F, Barwell L, Feyerabend S, Grande E, Martinez-Carrasco A, Font A, Berruti A, Sternberg CN, Jones R, Lefresne F, Lahaye M, Thomas S, Joshi S, Shen D, Ricci D, Gormley M, Merseburger AS, Tombal B, Annala M, Chi KN, De Giorgi U, Gonzalez-Billalabeitia E, Wyatt AW, Attard G. Plasma Androgen Receptor Copy Number Status at Emergence of Metastatic Castration-Resistant Prostate Cancer: A Pooled Multicohort Analysis. JCO Precis Oncol. 2019 Sep 24;3:PO.19.00123. doi: 10.1200/PO.19.00123. eCollection 2019. PMID 32923850
- [Derived] Attard G, Merseburger AS, Arlt W, Sternberg CN, Feyerabend S, Berruti A, Joniau S, Geczi L, Lefresne F, Lahaye M, Shelby FN, Pissart G, Chua S, Jones RJ, Tombal B. Assessment of the Safety of Glucocorticoid Regimens in Combination With Abiraterone Acetate for Metastatic Castration-Resistant Prostate Cancer: A Randomized, Open-label Phase 2 Study. JAMA Oncol. 2019 Aug 1;5(8):1159-1167. doi: 10.1001/jamaoncol.2019.1011. PMID 31246234

RESULTS

PARTICIPANT FLOW:
Groups:
- Abiraterone Acetate 1000 mg QD + Prednisone 5 mg BID: Participants received abiraterone acetate 1000 milligram (mg) tablet orally once daily (QD) and prednisone 5 mg tablet orally twice daily (BID) up to 156 Weeks. Participants who were progression-free at 156 weeks entered the extension phase of the study and received study treatment until death, radiographic disease progression and/or unequivocal clinical progression, and/or other specific reasons for discontinuation. Participants who ended the extension phase prematurely and participants who did not enter the extension phase entered a follow-up phase until end of study.
- Abiraterone Acetate 1000 mg QD + Prednisone 5 mg QD: Participants received abiraterone acetate 1000 mg and prednisone 5 mg tablet orally QD up to 156 Weeks. Participants who were progression-free at 156 weeks entered the extension phase of the study and received study treatment until death, radiographic disease progression and/or unequivocal clinical progression, and/or other specific reasons for discontinuation. Participants who ended the extension phase prematurely and participants who did not enter the extension phase entered a follow-up phase until end of study.
- Abiraterone Acetate 1000 mg QD + Prednisone 2.5 mg BID: Participants received abiraterone acetate 1000 mg tablet orally QD and prednisone 2.5 mg tablet orally BID up to 156 Weeks. Participants who were progression-free at 156 weeks entered the extension phase of the study and received study treatment until death, radiographic disease progression and/or unequivocal clinical progression, and/or other specific reasons for discontinuation. Participants who ended the extension phase prematurely and participants who did not enter the extension phase entered a follow-up phase until end of study.
- Abiraterone Acetate 1000 mg QD + Dexamethasone 0.5 mg QD: Participants received abiraterone acetate 1000 mg and dexamethasone 0.5 mg tablet orally QD up to 156 Weeks. Participants who were progression-free at 156 weeks entered the extension phase of the study and received study treatment until death, radiographic disease progression and/or unequivocal clinical progression, and/or other specific reasons for discontinuation. Participants who ended the extension phase prematurely and participants who did not enter the extension phase entered a follow-up phase until end of study.
Period: Overall Study
Arm/Group | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg BID | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg QD | Abiraterone Acetate 1000 mg QD + Prednisone 2.5 mg BID | Abiraterone Acetate 1000 mg QD + Dexamethasone 0.5 mg QD
Started | 41 | 41 | 40 | 42
Treated | 41 | 41 | 39 | 42
Completed | 0 | 0 | 0 | 0
Not Completed | 41 | 41 | 40 | 42
Not completed — Death | 25 | 15 | 27 | 20
Not completed — Lost to Follow-up | 3 | 4 | 3 | 2
Not completed — Withdrawal of consent | 2 | 5 | 1 | 2
Not completed — Study Terminated by Sponsor | 9 | 13 | 8 | 16
Not completed — Biochemical progression | 0 | 1 | 0 | 0
Not completed — Clinical progression | 0 | 0 | 1 | 0
Not completed — Disease progression | 1 | 0 | 0 | 0
Not completed — Patient decision | 0 | 0 | 0 | 1
Not completed — Patient to follow subsequent treatment | 0 | 1 | 0 | 0
Not completed — Progressive disease | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — PSA-progression | 0 | 1 | 0 | 0
Not completed — Study medication no longer effective | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg BID | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg QD | Abiraterone Acetate 1000 mg QD + Prednisone 2.5 mg BID | Abiraterone Acetate 1000 mg QD + Dexamethasone 0.5 mg QD | Total
Number analyzed (Participants) | 41 | 41 | 40 | 42 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (9.28) | 69 (8.44) | 69.3 (7.51) | 71.3 (8.12) | 69.6 (8.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 41 | 41 | 40 | 42 | 164
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 8 | 9 | 10 | 14 | 41
  Germany | 7 | 10 | 5 | 6 | 28
  United Kingdom | 10 | 9 | 8 | 8 | 35
  Hungary | 6 | 4 | 6 | 4 | 20
  Italy | 10 | 9 | 11 | 19 | 49

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Neither of the 2 Mineralocorticoid Excess Toxicity During the First 24 Weeks of Treatment
Description: No mineralocorticoid excess is defined as experiencing neither of the 2 mineralocorticoid excess toxicities, that is, neither hypokalemia nor hypertension.
Time Frame: Week 24
Population: Safety population included all randomized and treated participants. Here "N" (Number of Participants Analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg BID | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg QD | Abiraterone Acetate 1000 mg QD + Prednisone 2.5 mg BID | Abiraterone Acetate 1000 mg QD + Dexamethasone 0.5 mg QD
Number analyzed (Participants) | 34 | 38 | 35 | 37
Percentage of Participants | 70.6 [53.8 to 83.2] | 36.8 [23.4 to 52.7] | 60.0 [43.6 to 74.4] | 70.3 [54.2 to 82.5]

2. Secondary Outcome: Percentage of Participants With Confirmed Prostate Specific Antigen (PSA) Response Rate [Greater Than or Equal to (>=) 50 Percent (%) Decline From Baseline] at Week 12
Description: The PSA response is defined as a >= 50% decline from baseline according to the adapted Prostate Cancer Working Group 2 (PCWG2) criteria. For a PSA response to be confirmed, an additional PSA measurement obtained 4 or more weeks later has to show >=50% decline from baseline.
Time Frame: Week 12
Population: Intent-to-treat (ITT) population included all randomized participants regardless of whether they received any study treatment. Here "N" (Number of Participants Analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg BID | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg QD | Abiraterone Acetate 1000 mg QD + Prednisone 2.5 mg BID | Abiraterone Acetate 1000 mg QD + Dexamethasone 0.5 mg QD
Number analyzed (Participants) | 35 | 34 | 36 | 39
Percentage of Participants | 57.1 [40.9 to 72.0] | 70.6 [53.8 to 83.2] | 47.2 [32.0 to 63.0] | 79.5 [64.5 to 89.2]

3. Secondary Outcome: Change From Baseline to Endpoint in Brief Pain Inventory- Short Form (BPI-SF) Score: Worst Pain
Description: BPI-SF is 11-item self-reported questionnaire designed to assess severity and impact of pain on daily functions (pain interference). It includes 4 questions that assess pain intensity/severity (worst, least, average, right now) and 7 questions that assess impact of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life). BPI-SF scores range from 0=No pain to 10=Pain as bad as you can imagine; Higher scores indicate greater pain. Worst pain item has a scale of 0 to 10 with 0 indicating "No pain" and 10 indicating "Pain as bad as you can imagine". Last observation carried forward (LOCF) approach used for endpoint analysis. Last observation defined as last visit with non-missing data for parameter analyzed.
Time Frame: Baseline up to the Endpoint (last post-baseline assessment value during 156 weeks of main study treatment period [MSTP])
Population: ITT population included all randomized participants regardless of whether they received any study treatment. Here "N" (Number of Participants Analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg BID | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg QD | Abiraterone Acetate 1000 mg QD + Prednisone 2.5 mg BID | Abiraterone Acetate 1000 mg QD + Dexamethasone 0.5 mg QD
Number analyzed (Participants) | 36 | 33 | 37 | 38
Units on a scale | 1.6 (2.43) | 2.2 (2.86) | 2.5 (2.39) | 1.3 (2.28)

4. Secondary Outcome: Change From Baseline to Endpoint in Brief Pain Inventory- Short Form (BPI-SF) Score: Pain Intensity Subscale
Description: BPI-SF is 11-item self-reported questionnaire designed to assess severity and impact of pain on daily functions (pain interference). It includes 4 questions that assess pain intensity/severity (worst, least, average, right now) and 7 questions that assess impact of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life). BPI-SF scores range from 0=No pain to 10=Pain as bad as you can imagine; Higher scores indicate greater pain. Pain Severity Index is the mean of the 4 pain scores (worst, least, average, and right now) on the BPI-SF; range is 0=No pain to 10=Pain as bad as you can imagine; A higher score indicates greater pain severity. LOCF approach used for endpoint analysis. Last observation is defined as last visit with non-missing data for parameter analyzed.
Time Frame: Baseline up to the Endpoint (last post-baseline assessment value during 156 weeks of MSTP)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg BID | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg QD | Abiraterone Acetate 1000 mg QD + Prednisone 2.5 mg BID | Abiraterone Acetate 1000 mg QD + Dexamethasone 0.5 mg QD
Number analyzed (Participants) | 37 | 35 | 37 | 38
Units on a scale | 1.31 (1.788) | 1.37 (1.952) | 1.80 (2.014) | 0.97 (1.610)

5. Secondary Outcome: Change From Baseline to Endpoint in Brief Pain Inventory- Short Form (BPI-SF) Score: Pain Interference Subscale
Description: BPI-SF is 11-item self-reported questionnaire designed to assess severity and impact of pain on daily functions (pain interference). It includes 4 questions that assess pain intensity/severity (worst, least, average, right now) and 7 questions that assess impact of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life). BPI-SF scores range from 0=No pain to 10=Pain as bad as you can imagine; Higher scores indicate greater pain. Pain Interference Index is the mean of the scores for the 7 items of the BPI-SF; range is 0=Does not interfere to 10=Completely interferes. LOCF approach used for endpoint analysis. Last observation is defined as last visit with non-missing data for parameter analyzed.
Time Frame: Baseline up to the Endpoint (last post-baseline assessment value during 156 weeks of MSTP)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg BID | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg QD | Abiraterone Acetate 1000 mg QD + Prednisone 2.5 mg BID | Abiraterone Acetate 1000 mg QD + Dexamethasone 0.5 mg QD
Number analyzed (Participants) | 32 | 30 | 35 | 37
Units on a scale | 0.89 (1.794) | 1.76 (2.100) | 1.52 (2.180) | 1.12 (1.687)

6. Secondary Outcome: Change From Baseline to Endpoint in EuroQol-5 Dimension-5 Level (EQ-5D-5L): Index Score
Description: EQ-5D-5L measures health outcome self-completed by respondents. It consists of EQ-5D-5L descriptive system and EQ visual analogue scale (EQ-VAS). The descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each has 5 levels (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). Participant selects answer for each of 5 dimensions considering response that best matches his/her health "today". Responses were used to generate a Health Status Index (HSI). HSI ranges from -0.148 to 0.949 and is anchored at 0 (health state value equal to dead) and 1 (full health). LOCF approach used for endpoint analysis. Last observation is defined as last visit with non-missing data for parameter analyzed.
Time Frame: Baseline up to the Endpoint (last post-baseline assessment value during 156 weeks of MSTP)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg BID | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg QD | Abiraterone Acetate 1000 mg QD + Prednisone 2.5 mg BID | Abiraterone Acetate 1000 mg QD + Dexamethasone 0.5 mg QD
Number analyzed (Participants) | 37 | 38 | 36 | 38
Units on a scale | -0.0694 (0.18402) | -0.0638 (0.17772) | -0.0728 (0.18113) | -0.0359 (0.13515)

7. Secondary Outcome: Change From Baseline to Endpoint in EuroQol-5 Dimension-5 Level (EQ-5D-5L): EQ-VAS
Description: EQ-5D-5L measures health outcome self-completed by respondents. It consists of EQ-5D-5L descriptive system and EQ visual analogue scale (EQ-VAS). EQ-VAS self-rating records the respondent's own assessment of his/her overall health status at time of completion, on scale of 0 (the worst health you can imagine) to 100 (the best health you can imagine). LOCF approach used for endpoint analysis. Last observation is defined as last visit with non-missing data for parameter analyzed.
Time Frame: Baseline up to the Endpoint (last post-baseline assessment value during 156 weeks of MSTP)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg BID | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg QD | Abiraterone Acetate 1000 mg QD + Prednisone 2.5 mg BID | Abiraterone Acetate 1000 mg QD + Dexamethasone 0.5 mg QD
Number analyzed (Participants) | 38 | 37 | 37 | 37
Units on a scale | -4.5 (18.11) | -5.0 (16.82) | -6.6 (15.09) | -3.1 (13.00)

8. Secondary Outcome: Change From Baseline to Endpoint in Functional Assessment of Cancer Therapy-Prostate (FACT-P) Questionnaire Score
Description: FACT-P is a 39-item participant rated questionnaire which consists of 5 subscales assessing physical well-being (7 items; score range 0-28), social/family well-being (7 items; score range 0-28), emotional well-being (6 items; score range 0-24), functional well-being (7 items; score range 0-28), prostate-specific concerns (12 items; score range 0-48). Each item rated on 0 to 4 Likert type scale, then combined to produce subscale scores for each domain, as well as global quality of life (QoL) score that ranges from 0 to 156. Higher scores represent better QoL. Additional Concerns subscale has 12 items, each with a score 0-6 making a total subscale range 0-72 (higher scores are better). Missing data imputed as per FACT-P Ver4 scoring system (sum of item scores*number of items in subscale/number of items answered).
Time Frame: Baseline up to the Endpoint (last post-baseline assessment value during 156 weeks of MSTP)
Population: ITT population included all randomized participants regardless of whether they received any study treatment. Here,'n'(number of participants analyzed) signifies the number of participants analyzed in specific category.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg BID | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg QD | Abiraterone Acetate 1000 mg QD + Prednisone 2.5 mg BID | Abiraterone Acetate 1000 mg QD + Dexamethasone 0.5 mg QD
Number analyzed (Participants) | 41 | 41 | 40 | 42
Units on a scale
  Physical Well-Being: number analyzed (Participants) | 37 | 38 | 37 | 38
  Physical Well-Being | -0.98 (3.930) | -2.20 (4.449) | -2.46 (4.124) | -1.04 (3.268)
  Social/Family Well-Being: number analyzed (Participants) | 37 | 37 | 36 | 38
  Social/Family Well-Being | -0.01 (3.679) | 0.61 (3.794) | -0.78 (5.177) | -1.97 (5.749)
  Emotional Well-Being: number analyzed (Participants) | 37 | 38 | 35 | 36
  Emotional Well-Being | -1.46 (4.785) | -0.89 (3.289) | -1.66 (3.915) | -0.02 (3.542)
  Functional Well-Being: number analyzed (Participants) | 36 | 38 | 36 | 36
  Functional Well-Being | -1.13 (4.575) | -2.19 (5.767) | -2.67 (5.957) | -2.95 (6.698)
  Global Score: number analyzed (Participants) | 35 | 38 | 36 | 34
  Global Score | -4.73 (18.248) | -6.62 (17.118) | -10.39 (20.798) | -5.77 (18.322)
  Additional Concerns: number analyzed (Participants) | 37 | 38 | 37 | 38
  Additional Concerns | -1.29 (7.694) | -2.35 (6.342) | -3.96 (6.492) | -0.72 (6.080)

9. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS: Time from randomization to one of following: radiographic progression (RP), clinical progression (CP) or death. RP- per PCWG2 criteria and modified RECIST as time from randomization to one of following: 1) considered to have progressed by bone scan if: a) first scan with >=2 new lesions compared to baseline at <12 weeks from randomization and confirmed by second scan >=6 weeks later with >=2 additional new lesions, b) first scan with >=2 new lesions compared to baseline at >=12 weeks from randomization and new lesions on next bone scan >=6 weeks later; 2) Progression of soft tissue lesions per modified RECIST; CP: cancer pain requiring initiation of chronic use of opiate analgesia (oral use for >=3 weeks; parenteral use for >=7 days), Or immediate need to initiate cytotoxic chemotherapy or either radiation therapy or surgical intervention for complications due to tumor progression, even in absence of RP, Or deterioration in ECOG performance status to grade 3 or above.
Time Frame: Up to 4.9 years
Population: Efficacy analysis set included ITT population- all randomized participants regardless of whether they received any study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg BID | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg QD | Abiraterone Acetate 1000 mg QD + Prednisone 2.5 mg BID | Abiraterone Acetate 1000 mg QD + Dexamethasone 0.5 mg QD
Number analyzed (Participants) | 41 | 41 | 40 | 42
Months | 16.16 [9.95 to 23.75] | 12.68 [7.66 to 29.47] | 8.51 [5.62 to 15.44] | 21.22 [15.08 to 38.44]

10. Secondary Outcome: Time to Prostate-Specific Antigen (PSA) Progression
Description: Time to PSA progression was defined as time interval from the date of randomization to the date of the first prostate-specific antigen (PSA) progression as defined in the protocol-specific Prostate Specific Antigen Working Group 2 (PSAWG2) criteria during the main study treatment period. PCWG2 defines PSA progression as the date that a 25 percent (%) or greater increase and an absolute increase of 2 nanogram per milliliter (ng/mL) or more from the nadir is documented, which is confirmed by a second value obtained 3 or more weeks later.
Time Frame: Up to 156 weeks
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg BID | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg QD | Abiraterone Acetate 1000 mg QD + Prednisone 2.5 mg BID | Abiraterone Acetate 1000 mg QD + Dexamethasone 0.5 mg QD
Number analyzed (Participants) | 41 | 41 | 40 | 42
Months | 10.38 [10.05 to 20.99] | 10.22 [7.39 to 26.84] | 4.83 [2.79 to 10.15] | 18.56 [10.15 to NA] — Here 'NA' represents that upper limit of 95% Confidence Interval (CI) was not estimable due to a limited number of events and the small sample size.

11. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with measurable disease at baseline achieving a complete response (CR) or partial response (PR) according to modified response evaluation criteria in solid tumors (RECIST) criteria. RECIST criteria for CR: disappearance of all target lesions and non-target lesions , any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 millimetre [mm] short axis). PR: At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 4.9 years
Population: Efficacy analysis set included ITT population- all randomized participants regardless of whether they received any study treatment. Population included participants with measurable disease at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg BID | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg QD | Abiraterone Acetate 1000 mg QD + Prednisone 2.5 mg BID | Abiraterone Acetate 1000 mg QD + Dexamethasone 0.5 mg QD
Number analyzed (Participants) | 19 | 18 | 10 | 16
Percentage of participants | 42.1 | 38.9 | 60.0 | 56.3

12. Secondary Outcome: Time to Opiate Use for Cancer-related Pain
Description: Time to opiate use for cancer-related pain is defined the time interval from the date of randomization to the first date of opiate use for cancer pain.
Time Frame: Up to 156 weeks
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg BID | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg QD | Abiraterone Acetate 1000 mg QD + Prednisone 2.5 mg BID | Abiraterone Acetate 1000 mg QD + Dexamethasone 0.5 mg QD
Number analyzed (Participants) | 41 | 41 | 40 | 42
Months | NA [NA to NA] — Here "NA (not available)" signifies that median and 95% Confidence Interval (CI) were not estimable due to a limited number of events and the small sample size. | NA [NA to NA] — Here "NA (not available)" signifies that median and 95% Confidence Interval (CI) were not estimable due to a limited number of events and the small sample size. | NA [NA to NA] — Here "NA (not available)" signifies that median and 95% Confidence Interval (CI) were not estimable due to a limited number of events and the small sample size. | NA [NA to NA] — Here "NA (not available)" signifies that median and 95% Confidence Interval (CI) were not estimable due to a limited number of events and the small sample size.

13. Secondary Outcome: Time to Deterioration in Eastern Cooperative Oncology Group (ECOG) Performance Score by 1 Point
Description: Time to deterioration in ECOG Performance Status, the time interval from the date of randomization to the first date in which at least one point change (worsening) in the ECOG is observed during the main study treatment period. The ECOG performance status is a grade scale to measure quality of life (QoL). Scores run from 0 to 5, with 0 denoting perfect health and 5 denoting death.
Time Frame: Up to 156 weeks
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg BID | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg QD | Abiraterone Acetate 1000 mg QD + Prednisone 2.5 mg BID | Abiraterone Acetate 1000 mg QD + Dexamethasone 0.5 mg QD
Number analyzed (Participants) | 41 | 41 | 40 | 42
Months | NA [NA to NA] — Here 'NA' (not available)" signifies that median and 95% Confidence Interval (CI) were not estimable due to a limited number of events and the small sample size. | NA [NA to NA] — Here 'NA' (not available)" signifies that median and 95% Confidence Interval (CI) were not estimable due to a limited number of events and the small sample size. | NA [NA to NA] — Here 'NA' (not available)" signifies that median and 95% Confidence Interval (CI) were not estimable due to a limited number of events and the small sample size. | NA [23.95 to NA] — Here 'NA' (not available)" signifies that median and upper limit of 95% Confidence Interval (CI) were not estimable due to a limited number of events and the small sample size.

14. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time interval from the date of randomization to the date of death from any cause.
Time Frame: Up to 156 weeks
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg BID | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg QD | Abiraterone Acetate 1000 mg QD + Prednisone 2.5 mg BID | Abiraterone Acetate 1000 mg QD + Dexamethasone 0.5 mg QD
Number analyzed (Participants) | 41 | 41 | 40 | 42
Months | 34.07 [26.38 to 48.49] | 48.43 [39.95 to NA] — Here 'NA' (not available) signifies that upper limit of 95% Confidence Interval (CI) was not estimable due to a limited number of events and the small sample size. | 27.96 [23.66 to 40.51] | 42.81 [30.23 to NA] — Here 'NA' (not available) signifies that upper limit of 95% Confidence Interval (CI) was not estimable due to a limited number of events and the small sample size.

15. Secondary Outcome: Time to Next Prostate Cancer Therapy
Description: Time to next prostate cancer therapy is defined as the time interval from the date of randomization to the date of initiation of first next therapy for prostate cancer.
Time Frame: Up to 4.9 years
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg BID | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg QD | Abiraterone Acetate 1000 mg QD + Prednisone 2.5 mg BID | Abiraterone Acetate 1000 mg QD + Dexamethasone 0.5 mg QD
Number analyzed (Participants) | 41 | 41 | 40 | 42
Months | 20.14 [13.27 to 26.91] | 19.48 [12.09 to 33.08] | 16.66 [9.26 to 22.47] | 28.29 [20.83 to 38.90]

ADVERSE EVENTS:
Time Frame: Up to 4.9 years
Description: Safety population included all randomized and treated participants.
Arm/Group | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg BID | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg QD | Abiraterone Acetate 1000 mg QD + Prednisone 2.5 mg BID | Abiraterone Acetate 1000 mg QD + Dexamethasone 0.5 mg QD
Serious Adverse Events (participants affected / at risk) | 12/41 | 10/41 | 11/39 | 18/42
Other Adverse Events (participants affected / at risk) | 39/41 | 36/41 | 37/39 | 39/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg BID (N=41) | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg QD (N=41) | Abiraterone Acetate 1000 mg QD + Prednisone 2.5 mg BID (N=39) | Abiraterone Acetate 1000 mg QD + Dexamethasone 0.5 mg QD (N=42)
Anaemia of Malignant Disease (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Atrial Flutter (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac Failure (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 1 | 0 | 0
Device Occlusion (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Neuroendocrine Carcinoma of the Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Dizziness Postural (Nervous system disorders) | 0 | 0 | 0 | 1
Hypokinesia (Nervous system disorders) | 0 | 0 | 1 | 0
Nerve Root Compression (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1
Bladder Tamponade (Renal and urinary disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0
Anaemia of Malignant Disease (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Atrial Flutter (Cardiac disorders) | 0 | 1 | 0 | 0
Atrioventricular Block Second Degree (Cardiac disorders) | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac Failure (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Incarcerated Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Obstructive Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatic Cyst (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Death (General disorders) | 0 | 1 | 0 | 0
General Physical Health Deterioration (General disorders) | 1 | 0 | 0 | 0
Performance Status Decreased (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 2
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Ketosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Neuroendocrine Carcinoma of the Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Dementia Alzheimer's Type (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness Postural (Nervous system disorders) | 0 | 0 | 0 | 1
Frontotemporal Dementia (Nervous system disorders) | 0 | 0 | 0 | 1
Haemorrhage Intracranial (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Hypokinesia (Nervous system disorders) | 0 | 0 | 1 | 0
Nerve Root Compression (Nervous system disorders) | 0 | 0 | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 2 | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 1 | 3
Device Occlusion (Product Issues) | 1 | 0 | 0 | 0
Psychotic Disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1 | 0 | 1
Bladder Tamponade (Renal and urinary disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 2
Renal Colic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 1
Pelvic Pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Circulatory Collapse (Vascular disorders) | 0 | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg BID (N=41) | Abiraterone Acetate 1000 mg QD + Prednisone 5 mg QD (N=41) | Abiraterone Acetate 1000 mg QD + Prednisone 2.5 mg BID (N=39) | Abiraterone Acetate 1000 mg QD + Dexamethasone 0.5 mg QD (N=42)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 1
Abdominal Pain (Gastrointestinal disorders) | 4 | 1 | 4 | 1
Constipation (Gastrointestinal disorders) | 6 | 2 | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 1
Asthenia (General disorders) | 2 | 3 | 1 | 1
Fatigue (General disorders) | 1 | 6 | 4 | 4
Oedema Peripheral (General disorders) | 6 | 4 | 2 | 4
Pyrexia (General disorders) | 1 | 0 | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2 | 2
Alanine Aminotransferase Increased (Investigations) | 1 | 2 | 3 | 4
Aspartate Aminotransferase Increased (Investigations) | 0 | 2 | 3 | 3
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 1 | 1 | 3
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 0 | 2 | 0
C-Reactive Protein Increased (Investigations) | 0 | 0 | 2 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 6 | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4 | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 8 | 4
Bone Pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 3 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2
Headache (Nervous system disorders) | 1 | 2 | 2 | 2
Haematuria (Renal and urinary disorders) | 1 | 1 | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 3 | 1
Hot Flush (Vascular disorders) | 2 | 1 | 1 | 3
Hypertension (Vascular disorders) | 6 | 15 | 12 | 5
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 4
Abdominal Pain (Gastrointestinal disorders) | 4 | 2 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 1 | 3 | 2
Constipation (Gastrointestinal disorders) | 9 | 4 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 2 | 1
Dry Mouth (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 2 | 3
Vomiting (Gastrointestinal disorders) | 2 | 2 | 2 | 2
Asthenia (General disorders) | 3 | 4 | 1 | 1
Chest Pain (General disorders) | 0 | 3 | 1 | 1
Fatigue (General disorders) | 2 | 6 | 5 | 7
Influenza Like Illness (General disorders) | 3 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 8 | 4 | 4 | 8
Pyrexia (General disorders) | 1 | 1 | 2 | 1
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 3
Nasopharyngitis (Infections and infestations) | 3 | 1 | 3 | 2
Urinary Tract Infection (Infections and infestations) | 1 | 4 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 2
Alanine Aminotransferase Increased (Investigations) | 3 | 2 | 3 | 5
Aspartate Aminotransferase Increased (Investigations) | 1 | 2 | 3 | 4
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 1 | 1 | 3
Blood Bilirubin Increased (Investigations) | 3 | 0 | 1 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 0 | 2 | 0
C-Reactive Protein Increased (Investigations) | 0 | 0 | 2 | 0
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 0 | 3
Weight Decreased (Investigations) | 7 | 7 | 10 | 3
Weight Increased (Investigations) | 4 | 2 | 1 | 6
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 1 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 7 | 7 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 9 | 2 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 13 | 5 | 10 | 9
Bone Pain (Musculoskeletal and connective tissue disorders) | 11 | 3 | 5 | 2
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 | 1 | 4 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 | 2 | 4 | 3
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 2 | 3
Paraesthesia (Nervous system disorders) | 0 | 0 | 2 | 2
Haematuria (Renal and urinary disorders) | 2 | 1 | 2 | 3
Urinary Retention (Renal and urinary disorders) | 2 | 3 | 0 | 1
Pelvic Pain (Reproductive system and breast disorders) | 3 | 2 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 3 | 1
Skin Atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3
Hot Flush (Vascular disorders) | 3 | 1 | 3 | 5
Hypertension (Vascular disorders) | 14 | 22 | 13 | 10

LIMITATIONS AND CAVEATS:
Study not designed/powered to allow comparisons in study groups. Per protocol amendment 6, the study was ended earlier since sufficient extension and follow-up data have been collected to allow statistical analysis of secondary objectives.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.